CLINICAL TRIAL: NCT04091269
Title: Automatic Adjustmen of Inspiratory Triger and Cycling-off Based on Waveform Improved Patient-ventilator Interation During Pressure Support Ventilation
Brief Title: IntelliCycleTM 2.0 Improved Patient-ventilator Asynchrony During PSV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Principal Investigator, Southeast University, China
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ZDSYLL067-P01
Record Dates: First submitted 2019-09-11; First posted 2019-09-16 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Automatic Adjustmen of Inspiratory Triger and Cycling-off
Keywords: patient-ventilator interation; automatic adjustmen of inspiratory triger and cycling-off; Neurally controlled PS

STUDY DESIGN:
Intervention Model Description: PSV+ Automatic adjustmen of inspiratory triger and cycling-off based on waveform PSV with fixed inspiratory and expiratory NAVA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- PSV-10% (Placebo Comparator): PSV mode using E5 ventilator with fixed flow trigger and Esense 10%
  Interventions: Device: automatic adjustmen of inspiratory triger and cycling-off based on waveform and PSV with fixed Esence
- PVS-30% (Placebo Comparator): PSV mode using E5 ventilator with fixed flow trigger and Esense 30%
  Interventions: Device: automatic adjustmen of inspiratory triger and cycling-off based on waveform and PSV with fixed Esence
- PSV-50% (Placebo Comparator): PSV mode using E5 ventilator with fixed flow trigger and Esense 50%
  Interventions: Device: automatic adjustmen of inspiratory triger and cycling-off based on waveform and PSV with fixed Esence
- PSV-auto (Experimental): PSV mode using automatic adjustmen of inspiratory triger and cycling-off based on waveform
  Interventions: Device: automatic adjustmen of inspiratory triger and cycling-off based on waveform and PSV with fixed Esence
- PSV-neuro (Active Comparator): NAVA mode using NAVA level of 15 cmH2O/uV and pressure limit function to simulated EAdi triggered PSV.
  Interventions: Device: automatic adjustmen of inspiratory triger and cycling-off based on waveform and PSV with fixed Esence

INTERVENTIONS:
Device: automatic adjustmen of inspiratory triger and cycling-off based on waveform and PSV with fixed Esence — The ventilators have a compunter drived funcation of automatic adjustmen of inspiratory triger and cycling-off based on waveform, IntelliCycleTM 2.0.

SUMMARY:
Pressure Support Ventilation use Expiratory triggering sensitivity (Esense) to transfer inspiration to expiration, the value of Esense is fixed. That may lead to asynchrony between humans and ventilators, making people uncomfortable and prolonging weaning time. Furthermore，trigger delay or inffective trigger happens frequently during insppiratory triggering. The ventilators have a compunter drived funcation of automatic adjustmen of inspiratory triger and cycling-off based on waveform, IntelliCycleTM 2.0. It will make the transforming more synchrony with humans. The objectibe of the present study is to detect the effect of automatic adjustmen of inspiratory triger and cycling-off based on waveform on patient-ventilator interation.

DETAILED DESCRIPTION:
This is a physiological cross-over study. Enrolled patient with different baseline respiratory mechanics, for example ARDS patients with low compliance, COPD patient with high airway resistance and postoperative patients with almost normal compliance and airway resistance. Patients are ventilated with PSV+ Automatic adjustmen of inspiratory triger and cycling-off based on waveform, PSV with fixed inspiratory and expiratory and NAVA in two different levels of support. The demographic characteristics, diagnosis, formerly medical history, Ventilator indications, Ventilator data, other respiratory treatments, patient-ventilator interation, work of breathing, Eadi, will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Postoperation patients

1. receiving invasive mechanical ventilation due to operation
2. abdominal surgery, orthopedic surgery or gynecological surgery
3. without respiratory system Comorbidity
4. able to sustain PSV more than 1 h with inspiratory support ≤ 15 cmH2O.

COPD and ARDS patients

1. receiving invasive mechanical ventilation due to acute respiratory failure
2. able to sustain PSV more than 1 h with inspiratory support ≤ 15 cmH2O.

Exclusion Criteria:

1. age < 18 or >85 years,
2. tracheostomy at time of inclusion,
3. contra-indication for nasogastric tube insertion (e.g. history of esophageal varices, gastro-esophageal surgery in the previous 12 months or gastro-esophageal bleeding in the previous 7 days, INR ratio > 1.5 , APTT > 44 s, history of leukemia),
4. neuromuscular disease affecting spontaneous breathing (e.g. history of acute central or peripheral nervous system disorder or neuromuscular disease with irregular spontaneous rhythm),
5. hemodynamic unstable (heart rate > 140 beats/min, vasopressors required with ≥ 5 μg.kg-1.min-1 dopamine/ dobutamine, or ≥ 0.2 μg.kg-1.min-1 norepinephrine),
6. sedation level Richmond Agitation-Sedation Scale (RASS) ≤ -2 or ≥ 2,
7. lack of informed consent and patients included in other intervention study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Asynchrony Index | 20 minutes
  number of asynchrony events divided by the total neural respiratory rate

SECONDARY OUTCOMES:
Patient Respiratory Patterns | 20 minutes
  Patient Respiratory Patterns during Pressure Support Ventilation
gas exchange | 20 minutes
  Patient gas exchange during Pressure Support Ventilation
work of breathing | 20 minutes
  work of triggering and respiratory in different arms
other patient-ventilator synchrony parameters | 20minutes
  trigger and cycle-off asynchrony, Ineffective efforts, double triggering, auto-triggering, premature cycling and late cycling

CONTACTS AND LOCATIONS:
Overall Officials: Ling Liu, Study Director — Zhongda Hospital, School of Medicine, Southeast University,
Locations (1):
- Ling Liu, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided